CLINICAL TRIAL: NCT02368691
Title: A Phase 2 Open Label, Multi-Center, Multinational Study Investigating The Efficacy and Safety Of GTx-024 On Advanced, Androgen Receptor-Positive Triple Negative Breast Cancer (AR+ TNBC)
Brief Title: Efficacy and Safety of GTx-024 in Patients With Androgen Receptor-Positive Triple Negative Breast Cancer (AR+ TNBC)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of Efficacy
Sponsor: GTx (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G200901
Record Dates: First submitted 2015-02-10; First posted 2015-02-23 (Estimated); Results first posted 2020-10-30 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-10

CONDITIONS: Triple Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — ostarine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- GTx-024 (Experimental): GTx-024 capsules, 18 mg PO once-daily for up to 12 months
  Interventions: Drug: GTx-024

INTERVENTIONS:
Drug: GTx-024 — GTx-024 softgel capsules will be administered once-daily to a total dose of 18 mg
  Other Names: Enobosarm; Ostarine; S-22

SUMMARY:
The purpose of this study is to determine if GTx-024 is effective and safe in the treatment of patients with advanced, androgen receptor positive triple negative breast cancer (AR+ TNBC).

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to give voluntary, written and signed, informed consent
* Women ≥ 18 years of age
* Women with TNBC who have received at least one but no more than two prior chemotherapy regimens for TNBC
* Confirmation of AR+ (defined as ≥ 10% nuclear AR staining by immunohistochemistry [IHC]) TNBC in either the primary or metastatic lesion, assessed during the screening period by a local laboratory or by medical history
* TNBC confirmed by medical history as: human epidermal growth factor receptor 2 [HER2]-negative (confirmed by IHC 0, 1+ regardless of fluorescence in situ hybridization [FISH] ratio; IHC 2+ with FISH ratio lower than 2.0 or HER2 gene copy less than 6.0; FISH ratio of 0, indicating gene deletion, when positive and negative in situ hybridization [ISH] controls are present); estrogen receptor (ER) negative (confirmed as ER expression less than or equal to 1% positive tumor nuclei); progesterone receptor negative (confirmed as progesterone receptor expression less than or equal to 1% positive tumor nuclei)
* Availability of paraffin embedded or formalin fixed tumor tissue; OR, a minimum of 10 and up to 20 slides of archived tumor tissue for central laboratory confirmation of AR status and molecular subtyping. Metastatic tumor tissue is preferred when possible
* Subjects must have either measurable disease or bone-only non-measurable disease, evaluable according to RECIST 1.1
* Subjects with bone metastases should be treated with intravenous bisphosphonates or subcutaneous denosumab (or investigator preferred standard of care) prior to and during the trial, unless there is a contraindication or subject intolerance to these therapies
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1 at the time of screening and enrollment
* Negative pregnancy test in women of childbearing potential (premenopausal or less than 12 months of amenorrhea post-menopause, and who have not undergone surgical sterilization), no more than 7 days before the first dose of study treatment
* For women of childbearing potential who are sexually active, agreement to use a highly effective, non-hormonal form of contraception during and for at least 6 months after completion of study treatment; OR, a fertile male partner willing and able to use effective non-hormonal of contraception (barrier method of contraception in conjunction with spermicidal jelly, or surgical sterilization) during and for at least 6 months after completion of study treatment
* Adequate organ function as shown by:

  * Absolute neutrophil count ≥ 1,000 cells/mm3
  * Platelet count ≥ 100,000 cells/mm3
  * Hemoglobin ≥ 9 g/dL
  * Serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 Upper Limit of the Normal range (ULN) (or ≤ 5 if hepatic metastases are present)
  * Total serum bilirubin ≤ 2.0 × ULN (unless the subject has documented Gilbert Syndrome)
  * Alkaline phosphatase levels ≤ 2.5 × ULN (≤ 5 × ULN in subjects with liver metastasis)
  * Serum creatinine < 2.0 mg/dL or 177 μmol/L
  * International normalized ratio (INR), activated partial thromboplastin time (aPTT), or partial thromboplastin time (PTT) < 1.5 × ULN (unless on anticoagulant treatment at screening)
* Able to swallow capsules
* Any toxicity from prior chemotherapy has resolved or Grade 1 (NCI-CTCAE, Version 4.0)

Exclusion Criteria:

* Life expectancy < 4 months;
* Subjects with radiographic evidence of central nervous system (CNS) metastases as assessed by computerized tomography (CT) or magnetic resonance imaging (MRI) that are not well controlled (symptomatic or requiring control with continuous corticosteroid therapy [e.g., dexamethasone]). Note: Subjects with CNS metastases are permitted to participate in the study if the CNS metastases are medically well controlled prior to screening (as assessed by the Investigator) after receiving local therapy (irradiation, surgery, etc.)
* Radiotherapy within 14 days prior to first dose of study treatment
* Have, in the judgment of the Investigator, a clinically significant concurrent illness or psychological, familial, sociological, geographical, or other concomitant condition that would not permit adequate follow-up and compliance with the study protocol
* Positive hepatitis B virus (HBV) and/or hepatitis C virus (HCV) infection at screening
* Positive human immunodeficiency virus (HIV) infection at screening
* Prior treatment with any anti-androgens, including but not limited to, enzalutamide and bicalutamide
* Major surgery within 28 days of the first dose of study treatment
* Be currently taking or have previously taken testosterone, methyltestosterone, oxandrolone (Oxandrin®), oxymetholone, danazol, fluoxymesterone (Halotestin®), testosterone-like agents (such as dehydroepiandrosterone, androstenedione, and other androgenic compounds, including herbals), or anti-androgens
* Treatment with any of the following hormone replacement therapies, unless discontinued at least 14 days prior to the first dose of study treatment:

  * Estrogens
  * Megesterol acetate
* Treatment with any investigational agent within 28 days before the first dose of study treatment
* Another active cancer (excluding adequately treated basal cell carcinoma or cervical intraepithelial neoplasia [CIN]/cervical carcinoma in situ or melanoma in situ). Prior history of other cancer is allowed as long as there is no active disease within the prior 5 years
* Subject has a concomitant medical condition that precludes adequate study treatment compliance or assessment, or increases subject risk, in the opinion of the Investigator, such as but not limited to:

  * Myocardial infarction or arterial thromboembolic events within 6 months prior to baseline or severe or unstable angina, New York Heart Association (NYHA) Class III or IV disease, or a QTcB (corrected according to Bazett's formula) interval > 470 msec; serious uncontrolled cardiac arrhythmia grade II or higher according to NYHA; uncontrolled hypertension (systolic > 150 and/or diastolic > 100 mm Hg)
  * Acute and chronic active infectious disorders and non-malignant medical illnesses that are uncontrolled or whose control may be jeopardized by the complications of this study therapy
  * Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of study drugs (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome)
* Current treatment with intravenous bisphosphonate or denosumab with elevated serum calcium corrected for albumin or ionized calcium levels outside institutional normal limits at screening
* History of non-compliance to medical regimens
* Subjects unwilling to or unable to comply with the protocol procedures as assessed by the Investigator
* Concurrent participation in another therapeutic clinical trial

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2017-09-22 (Actual); Study Completion 2017-09-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hope S Rugo, MD, Principal Investigator — University of California, San Francisco
Locations (7):
- United States (7):
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Lakeland Regional Health Care/Cancer Center, Lakeland, Florida
  - University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - St. Vincent Frontier Cancer Center, Billings, Montana
  - The West Clinic, PC, Memphis, Tennessee
  - US Oncology / Texas Oncology, P.A., Houston, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Up to 55 patients were planned for enrollment
Pre-assignment Details: No patients were excluded from the study before drug assignment
Period: Overall Study
Arm/Group | GTx-024
Started | 32 (32 subjects were enrolled and received at least one dose of study drug)
Completed | 0
Not Completed | 32
Not completed — Death | 13
Not completed — Lack of Efficacy | 15
Not completed — Physician Decision | 4

BASELINE CHARACTERISTICS:
Arm/Group | GTx-024
Number analyzed (Participants) | 32
Age, Continuous [Median (Full Range); unit: years] | 65 [35 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 27
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 32
AR status-positive [Number; unit: participants] | 18

OUTCOME MEASURES:

1. Primary Outcome: Clinical Benefit Rate, in Centrally Confirmed Androgen Receptor Positive (AR+) Subjects
Description: To estimate the clinical benefit rate (defined as complete response, partial response, or stable disease) according to Response Evaluation Criteria in Solid Tumors v 1.1 (RECIST) as assessed by CT or MRI in subjects with centrally confirmed AR+ status. Clinical Benefit Rate=CR+PR+SD. Complete Response (CR), disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease, <30% decrease in sum of the longest diameter of target lesions.
Time Frame: Sixteen (16) weeks
Population: Subjects who were centrally confirmed as AR+
Measure: Count of Participants; unit: Participants
Arm/Group | GTx-024
Number analyzed (Participants) | 18
Participants | 1

2. Secondary Outcome: Clinical Benefit Rate, in Full Analysis Set
Description: To estimate the clinical benefit rate in all subjects who receive at least one dose of study medication (full analysis set), regardless of central confirmation of AR status.
Time Frame: Sixteen (16) weeks
Population: All subjects, regardless of AR status
Measure: Number; unit: participants
Arm/Group | GTx-024
Number analyzed (Participants) | 32
participants | 2

3. Secondary Outcome: Best Overall Response
Description: To assess best overall response as measured by RECIST 1.1 from the start of study treatment until the end of treatment taking into account any requirement for confirmation. Best overall response is reported as the best response (CR, PR or SD) by CT or MRI up through 11 months of treatment, median duration of treatment 1.9 months.
Time Frame: From treatment initiation to end of treatment (up through 11 months of treatment, median duration of treatment 1.9 months).
Measure: Number; unit: participants
Arm/Group | GTx-024
Number analyzed (Participants) | 32
participants | 6

4. Secondary Outcome: Progression Free Survival
Description: To assess progression free survival (PFS) defined as the time elapsed between initiation of treatment and tumor progression as measured by RECIST 1.1 or death.
Time Frame: From treatment initiation to tumor progression or death. PFS was assessed up to 11 months of treatment; median duration of treatment, 1.9 months
Population: All patients regardless of AR status
Measure: Number (95% Confidence Interval); unit: months
Arm/Group | GTx-024
Number analyzed (Participants) | 32
months | 1.9 [1.7 to 2.3]

5. Secondary Outcome: Time-to-progression
Description: To assess time to progression defined as time elapsed between treatment initiation and tumor progression as measured by RECIST 1.1 or death due to disease progression.
Time Frame: From treatment initiation to tumor progression or death. Time to progression was assessed up to 11 months of treatment; median duration of treatment, 1.9 months
Population: All subjects regardless of AR status
Measure: Number (95% Confidence Interval); unit: months
Arm/Group | GTx-024
Number analyzed (Participants) | 32
months | 1.9 [1.7 to 2.0]

6. Secondary Outcome: Duration of Response
Description: To assess the duration of response defined as the time from documentation of tumor response to disease progression or death
Time Frame: From time of documented tumor response to tumor progression or death. Duration of response was assessed through 11 months; median treatment duration, 1.9 months
Population: All subjects regardless of AR status
Measure: Median (Full Range); unit: months
Arm/Group | GTx-024
Number analyzed (Participants) | 32
months | 1.9 [0.1 to 11]

7. Secondary Outcome: Objective Response Rate
Description: To estimate the objective response rate (defined as complete response or partial response) according to RECIST 1.1.
Time Frame: Sixteen (16) weeks
Measure: Number; unit: participants
Arm/Group | GTx-024
Number analyzed (Participants) | 32
participants | 0

8. Other Pre Specified Outcome: Number of Participants With Adverse Events
Description: To describe the safety profile in subjects with TNBC and centrally confirmed AR+ as well as in all subjects enrolled and treated.
Time Frame: Up to twelve (12) months
Measure: Number; unit: participants
Arm/Group | GTx-024
Number analyzed (Participants) | 32
participants | 28

ADVERSE EVENTS:
Time Frame: one year
Arm/Group | GTx-024
All-Cause Mortality (participants affected / at risk) | 13/32
Serious Adverse Events (participants affected / at risk) | 5/32
Other Adverse Events (participants affected / at risk) | 28/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GTx-024 (N=32)
CHF (Cardiac disorders) | 1 (1)
pleural effusion (Cardiac disorders) | 1 (1)
pulmonary embolism (Vascular disorders) | 1 (1)
tumor flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
UTI (Renal and urinary disorders) | 1 (1)
dehydration (Metabolism and nutrition disorders) | 1 (1)
constipation (Gastrointestinal disorders) | 1 (1)
rib fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GTx-024 (N=32)
investigations (Investigations) | 13 (13)
GI (Gastrointestinal disorders) | 8 (8)
metabolism (Metabolism and nutrition disorders) | 8 (8)
blood disorder (Blood and lymphatic system disorders) | 4 (4)
nervous system (Nervous system disorders) | 3 (3)
rash (Skin and subcutaneous tissue disorders) | 3 (3)

LIMITATIONS AND CAVEATS:
Early termination due to lack of efficacy and limited data reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-26): https://cdn.clinicaltrials.gov/large-docs/91/NCT02368691/Prot_SAP_000.pdf